CLINICAL TRIAL: NCT03767140
Title: Efficacy of Acupuncture in Exercise Tolerance in Patients With COPD Controlled, Randomized, Double Blind Study
Brief Title: Efficacy of Acupuncture in Exercise Tolerance in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciências Biomédicas Abel Salazar (Other)
Responsible Party: Principal Investigator, Carla Manuela Loureiro Barros, Master student, Instituto de Ciências Biomédicas Abel Salazar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: acupuncture
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: The patients were randomized in two groups, one verum acupuncture, submitted to real acupuncture treatment, and the other sham acupuncture, treated with false acupuncture.
  The method used to randomized was flipping a coin, when got heads they went to verum group and when got tails they went to sham group.
Who Masked: Participant, Investigator
Masking Description: Patients didn´t know what kind of therapy they were submitted The acupuncturist was a nurse, able to do invasive procedures with no knowledge of Chinese Medicine, and totally blind in terms of the verum or sham acupuncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum acupucnture (Experimental): Real acupuncture treatment
  Interventions: Procedure: acupuncture
- sham acupuncture (Sham Comparator): False acupuncture treatment using not acupuncture points
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — The patients were randomized in two groups, one verum acupuncture, submitted to real acupuncture treatment, and the other sham acupuncture, treated with false acupuncture

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is nowadays the 4th cause of death in the world and it´s expected to become the 3rd cause of death in 2020 and the majority cause of morbidity. Besides that, in Portugal COPD patients become more dependents each day.

Acupuncture as a reflex therapy it´s carried out through a Traditional Chinese Medicine (TCM) diagnose that will allowed to identify the acupoints.

The investigators are interested in to assess acupuncture efficacy on physical exercise tolerance in COPD patients.An experimental, controlled, randomized, double blind study was done. Patients were recruited according TCM diagnose to optimize potential therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD III,IV;
* able to walk;
* Informed consent signed;
* stable medication during last 3 days
* exacerbation during 3 months;
* Chinese diagnose opening principle;
* blood pressure "90"180 mmhg/ "100mmhg; respiratory rate "10"30 cpm

Exclusion Criteria:

* smoker;
* metastasis;
* hepatic,
* renal or cardiovascular disease;
* pulmonary hypertension;
* COPD symptoms exacerbation during the therapy;
* previous acupuncture treatments;
* unstable vital signs;
* pulmonary rehabilitation in the last 6 months;
* needle phobia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
six minute walk test (6MWT) | 6 minutes
  distance walked (metres)

SECONDARY OUTCOMES:
Oxygen peripheral saturation (SPO2) | 6 minutes
  pulse oximeter
Rating of perceived exertion (Borg Scale) | 6 minutes
  during 6MWT
Blood pressure | 6 minutes
  measure at end of 6MWT
heart rate | 6 minutes
  at end of 6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greten, Doctor, Study Chair — Abel Salazar Institute of Biomedical Sciences, University of Porto
Locations (1):
- Carla Manuela Loureiro Barros, Marco de Canaveses, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No